CLINICAL TRIAL: NCT01575197
Title: Immunogenicity of the Human Rotavirus Vaccine (Rotarix™) at Varying Schedules, Doses, and Ages in Rural Ghana
Brief Title: Evaluation of the Human Rotavirus Vaccine at Varying Schedules and Doses in Rural Ghana
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Noguchi Memorial Institute for Medical Research (Other); Navrongo Health Research Center (Unknown); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GHANA-HRV-01; OPP1017334 (Other Grant/Funding Number: Bill and Melinda Gates Foundation)
Record Dates: First submitted 2012-04-06; First posted 2012-04-11 (Estimated); Results first posted 2015-06-01 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-04

CONDITIONS: Rotavirus Gastroenteritis
MeSH Terms: interventions — RIX4414 vaccine

ARMS (3):
- Rotavirus Vaccine at age 6 & 10 weeks (Active Comparator): Participants are provided with the Human Rotavirus Vaccine (HRV) at 6 & 10 weeks of age.
  Interventions: Biological: Human Rotavirus Vaccine
- Rotavirus vaccine at age 10 & 14 weeks (Experimental): Participants are provided with the Human Rotavirus Vaccine (HRV) at 10 & 14 weeks of age.
  Interventions: Biological: Human Rotavirus Vaccine
- Rotavirus vaccine at age 6,10,&14 weeks (Experimental): Participants are provided with the Human Rotavirus Vaccine (HRV) at 6, 10, & 14 weeks of age.
  Interventions: Biological: Human Rotavirus Vaccine

INTERVENTIONS:
Biological: Human Rotavirus Vaccine — Rotavirus vaccine will be administered concomitantly with other routine Expanded Programme on Immunization (EPI) vaccinations at 6 & 10 weeks of age, 10 & 14 weeks of age, or 6, 10, & 14 weeks of age, depending on study arm assignment.
  Other Names: Rotarix

SUMMARY:
The purpose of this study is to determine whether giving the Human Rotavirus Vaccine on alternate dosing schedules will enhance the immune response to the vaccine in a low-resource, high-burden country in Africa. Alternate dosing schedules studied include giving the 2-dose vaccine schedule at a slightly older age and giving an additional dose of the vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Between 42 and 55 days of age at the time of enrollment.
* Healthy infant free of chronic or serious medical condition as determined by history and physical examination at the time of study enrollment.
* Parents/guardians of each subject are able to understand and follow study procedures and agree to participate in the study by providing parental/guardian permission.

Exclusion Criteria:

* If child has previously had intussusception or abdominal surgery.
* Use of any immunosuppressive drugs or immunoglobulin and/or blood product use since birth or anticipated during study period.
* Current enrollment in any other intervention trial or use of any investigational drug or vaccine throughout the study period.
* Birthweight less than 2000 grams or gestation < 36 weeks, if this information is available.
* Any subject who reports plan to leave the study area before the completion of the study (i.e., relocation, migration, etc.).
* Another child living in the same compound is already enrolled in the trial (i.e., only one participant can be enrolled per compound).
* After the rotavirus vaccine is introduced into the routine EPI system in Navrongo: Another child in the compound is less than 16 weeks of age.
* The child has received rotavirus vaccine outside of this study.

Ages: 42 Days to 55 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 456 (Actual)
Dates: Start 2012-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Armah, PhD, Principal Investigator — Noguchi Memorial Institute for Medical Research
Locations (1):
- Navrongo Health Research Center, Navrongo, Upper East Region, Ghana

REFERENCES:
- [Derived] Armah G, Lewis KD, Cortese MM, Parashar UD, Ansah A, Gazley L, Victor JC, McNeal MM, Binka F, Steele AD. A Randomized, Controlled Trial of the Impact of Alternative Dosing Schedules on the Immune Response to Human Rotavirus Vaccine in Rural Ghanaian Infants. J Infect Dis. 2016 Jun 1;213(11):1678-85. doi: 10.1093/infdis/jiw023. Epub 2016 Jan 27. PMID 26823335

RESULTS

PARTICIPANT FLOW:
Groups:
- Rotavirus Vaccine at Age 6 & 10 Weeks: Human rotavirus vaccine (HRV) was administered concomitantly with other routine Expanded Programme on Immunization (EPI) vaccinations at 6 & 10 weeks of age.
- Rotavirus Vaccine at Age 10 & 14 Weeks: Human rotavirus vaccine (HRV) was administered concomitantly with other routine Expanded Programme on Immunization (EPI) vaccinations at 10 & 14 weeks of age.
- Rotavirus Vaccine at Age 6,10,&14 Weeks: Human rotavirus vaccine (HRV) was administered concomitantly with other routine Expanded Programme on Immunization (EPI) vaccinations at 6, 10, & 14 weeks of age.
Period: Overall Study
Arm/Group | Rotavirus Vaccine at Age 6 & 10 Weeks | Rotavirus Vaccine at Age 10 & 14 Weeks | Rotavirus Vaccine at Age 6,10,&14 Weeks
Started | 152 | 152 | 152
Completed | 149 | 143 | 146
Not Completed | 3 | 9 | 6
Not completed — Migration out of study area | 1 | 5 | 4
Not completed — SAE | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Protocol Violation | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled subjects who received at least one rotavirus vaccine dose and are IgA seronegative (< 20 U/mL) at 6 (Groups 1 and 3) or 10 (Group 2) weeks of age at baseline.
Groups:
- Rotavirus Vaccine at Age 6 & 10 Weeks: Human rotavirus vaccine was administered concomitantly with other routine EPI vaccinations at 6 & 10 weeks of age.
- Rotavirus Vaccine at Age 10 & 14 Weeks: Human rotavirus vaccine was administered concomitantly with other routine EPI vaccinations at 10 & 14 weeks of age.
- Rotavirus Vaccine at Age 6,10,&14 Weeks: Human rotavirus vaccine was administered concomitantly with other routine EPI vaccinations at 6, 10, & 14 weeks of age.
- Total: Total of all reporting groups
Arm/Group | Rotavirus Vaccine at Age 6 & 10 Weeks | Rotavirus Vaccine at Age 10 & 14 Weeks | Rotavirus Vaccine at Age 6,10,&14 Weeks | Total
Number analyzed (Participants) | 150 | 149 | 151 | 450
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 6.2 (0.2) | 6.2 (0.2) | 6.2 (0.2) | 6.2 (0.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 79 | 72 | 219
  Male | 82 | 70 | 79 | 231
Region of Enrollment [Number; unit: participants]
  Ghana | 150 | 149 | 151 | 450

OUTCOME MEASURES:

1. Primary Outcome: Immunoglobulin A (IgA) Seroconversion: 6 & 10 Week vs. 6, 10, & 14 Week Vaccination Schedules
Description: Anti-rotavirus IgA seroconversion will be defined as the detection of anti-rotavirus IgA antibodies at a concentration ≥20 U/mL post-vaccination in infants seronegative for anti-rotavirus IgA pre-vaccination as measured by Enzyme Immunoassay (EIA).
Time Frame: 4-weeks post-vaccination (All Groups) and 8 weeks post-vaccination (6 & 10 week Group)
Population: Per-protocol analysis population--participants who (1) meet inclusion/exclusion criteria; (2) seronegative pre- vaccination; (3) concomitant administration of HRV and oral polio vaccine (OPV) according to Group schedule, (4) study visits in window periods (vaccination visits 4 weeks + 2 weeks), and (5) valid serology results.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rotavirus Vaccine at Age 6 & 10 Weeks | Rotavirus Vaccine at Age 6,10,&14 Weeks
Number analyzed (Participants) | 142 | 143
percentage of participants | 28.9 [22.1 to 36.8] | 43.4 [35.5 to 51.6]
Statistical Analysis 1: Comparison: Rotavirus Vaccine at Age 6 & 10 Weeks vs Rotavirus Vaccine at Age 6,10,&14 Weeks; Test type: Superiority or Other; p = 0.014, Fisher Exact

2. Secondary Outcome: IgA Seroconversion: 6 & 10 Week vs. 10 & 14 Week Vaccination Schedules
Description: Anti-rotavirus IgA seroconversion will be defined as the detection of anti-rotavirus IgA antibodies at a concentration ≥20 U/mL post-vaccination in infants seronegative for anti-rotavirus IgA pre- vaccination as measured by EIA.
Time Frame: 4-weeks post-vaccination (All Groups) and 8 weeks post-vaccination (6 & 10 week Group)
Population: Per-protocol analysis population--participants who (1) meet inclusion/exclusion criteria; (2) seronegative pre- vaccination; (3) concomitant administration of HRV and OPV according to Group schedule, (4) study visits in window periods (vaccination visits 4 weeks + 2 weeks), and (5) valid serology results.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rotavirus Vaccine at Age 6 & 10 Weeks | Rotavirus Vaccine at Age 10 & 14 Weeks
Number analyzed (Participants) | 142 | 139
percentage of participants | 28.9 [22.1 to 36.8] | 37.4 [29.8 to 45.7]
Statistical Analysis 1: Comparison: Rotavirus Vaccine at Age 6 & 10 Weeks vs Rotavirus Vaccine at Age 10 & 14 Weeks; Test type: Superiority or Other; p = 0.16, Fisher Exact

3. Secondary Outcome: IgA Geometric Mean Titers (GMTs): 6 & 10 Week vs. 6, 10, & 14 Week Vaccination Schedules
Description: IgA GMTs measured by EIA will be compared post-vaccination between participants receiving Rotarix at 6 and 10 weeks of age and those receiving Rotarix at 6, 10, and 14 weeks of age. For participants in Group 1, where post-vaccination response was measured at both 14 and 18 weeks of age, the highest response between these two visits was used as the final response for comparison.
Time Frame: 4-weeks post-vaccination (All Groups) and 8 weeks post-vaccination (6 & 10 week Group)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Rotavirus Vaccine at Age 6 & 10 Weeks | Rotavirus Vaccine at Age 6,10,&14 Weeks
Number analyzed (Participants) | 142 | 143
titers | 22.5 [17.4 to 28.2] | 32.6 [24.7 to 43.2]
Statistical Analysis 1: Comparison: Rotavirus Vaccine at Age 6 & 10 Weeks vs Rotavirus Vaccine at Age 6,10,&14 Weeks; Test type: Superiority or Other; p = 0.038, t-test, 2 sided

4. Secondary Outcome: IgA GMTs: 6 & 10 Week vs. 10 & 14 Week Vaccination Schedule
Description: IgA GMTs measured by EIA will be compared post-vaccination between participants receiving Rotarix at 6 and 10 weeks of age and those receiving Rotarix at 10 and 14 weeks of age. For participants in Group 1, where post-vaccination response was measured at both 14 and 18 weeks of age, the highest response between these two visits was used as the final response for comparison.
Time Frame: 4-weeks post-vaccination (All Groups) and 8 weeks post-vaccination (6 & 10 week Group)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Rotavirus Vaccine at Age 6 & 10 Weeks | Rotavirus Vaccine at Age 10 & 14 Weeks
Number analyzed (Participants) | 142 | 139
titers | 22.1 [17.4 to 28.2] | 26.5 [20.7 to 34.0]
Statistical Analysis 1: Comparison: Rotavirus Vaccine at Age 6 & 10 Weeks vs Rotavirus Vaccine at Age 10 & 14 Weeks; Test type: Superiority or Other; p = 0.30, t-test, 2 sided

5. Secondary Outcome: Baseline Immunoglobulin G (IgG) Levels: Impact on IgA Seroconversion Post-vaccination
Description: The number and percentage of participants demonstrating IgA seroconversion post-vaccination as defined above in infants seronegative for anti-rotavirus IgA pre- vaccination using the EIA assay) by EIA pre- and post-vaccination will be compared between participants in each group who had low as compared to high rotavirus immunoglobulin G (IgG) antibody levels pre-vaccination (i.e., at 6 weeks in Groups 1 and 3 and at 10 weeks in Group 2) as measured by Enzyme linked immunosorbent assay (ELISA). Low and high IgG categories will be determined based on the IgG antibody level distribution.
Time Frame: Baseline, 4-weeks post-vaccination (All Groups) and 8 weeks post-vaccination (6 & 10 week Group)
Reporting Status: Not Posted

6. Secondary Outcome: Vaccine-type Rotavirus Shedding in Stool
Description: Vaccine-type rotavirus shedding in the stool at 4 (±1 day) and 7 days (±1 day) following each Rotarix vaccination will be identified using EIA for rotavirus antigens and compared to baseline levels obtained just prior to each study vaccination. If shedding in stool is detected at either time point (per manufacturer's specifications) following each Rotarix vaccination, this will be considered evidence of vaccine take.
Time Frame: Days 4 and 7 post each study vaccination
Reporting Status: Not Posted

7. Secondary Outcome: SAE Assessment
Description: Serious adverse events (SAEs) occurring at anytime during the study will be measured as observed by study staff and/or reported by parent at any time. SAEs will be subcategorized according to treatment group as those deemed related to vaccination or not by an independent study monitor.
Time Frame: Throughout study period; Group 1: from enrollment through approximately 8 weeks of study participation, Groups 2 & 3: from enrollment through approximately 12 weeks of study participation
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events: 1 month following each study vaccination; serious adverse events: throughout study period, up to 5 months
Description: Any participant receiving one or more doses of rotavirus vaccine was included in this analysis.
Arm/Group | Rotavirus Vaccine at Age 6 & 10 Weeks | Rotavirus Vaccine at Age 10 & 14 Weeks | Rotavirus Vaccine at Age 6,10,&14 Weeks
Serious Adverse Events (participants affected / at risk) | 1/152 | 4/152 | 3/151
Other Adverse Events (participants affected / at risk) | 78/152 | 76/152 | 71/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotavirus Vaccine at Age 6 & 10 Weeks (N=152) | Rotavirus Vaccine at Age 10 & 14 Weeks (N=152) | Rotavirus Vaccine at Age 6,10,&14 Weeks (N=151)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abscess of the Left Jaw (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute Respiratory Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Congenital Hydrocephalus (Congenital, familial and genetic disorders) | 0 (0) | 1 (2) | 0 (0)
Gluteal Abscess/ Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotavirus Vaccine at Age 6 & 10 Weeks (N=152) | Rotavirus Vaccine at Age 10 & 14 Weeks (N=152) | Rotavirus Vaccine at Age 6,10,&14 Weeks (N=151)
Abdominal Pain/Diarrhea (Gastrointestinal disorders) | 27 (27) | 37 (37) | 27 (27)
Infection/Abscess/Boil/Sepsis (Infections and infestations) | 29 (29) | 25 (25) | 26 (26)
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 44 (44) | 45 (45) | 43 (43)
Fever (Infections and infestations) | 10 (10) | 7 (7) | 0 (0)
Malaria (Infections and infestations) | 14 (14) | 15 (15) | 12 (12)
Otitis Media (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Irritable/refusing to feed (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less